CLINICAL TRIAL: NCT03568253
Title: Longitudinal Follow-up of High Viscosity Glassionomer IonoStar Plus Versus a Composite Bulk X-tra-Fil Combined With Futurabond U (Splith Mouth Study)
Brief Title: Longitudinal Follow-up of High Viscosity Glassionomer IonoStar Plus Versus a Composite Bulk X-tra-Fil Combined With Futurabond U (Splith Mouth Study): Reunion Island, Circus of Mafate
Acronym: CVB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid situation / recruitment difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7550
Record Dates: First submitted 2018-05-14; First posted 2018-06-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Caries
Keywords: Bulk composite; High viscisity glassionomer; Cambra application (Caries management by risk assessment); E-dentistry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulk fil composite (Active Comparator)
  Interventions: Other: Caries treatment
- High viscosity glass ionomer (Active Comparator)
  Interventions: Other: Caries treatment

INTERVENTIONS:
Other: Caries treatment — Treatment by Bulk fil composite after randomization of the tooth
  Arms: Bulk fil composite
Other: Caries treatment — Treatment by High viscosity glass ionomer after randomization of the tooth
  Arms: High viscosity glass ionomer

SUMMARY:
The main objective is the longitudinal follow-up and comparison of the maintenance of the dental filling materials up to 24 months using the HVGIC IonoStar Plus versus Bulk X-Tra -Fil composite (Futurabond U adhesive system). 150 patients will be recruited in the Mafate dental health center. Patients with minimum 2 carious lesions (or multiple of 2, maximum 6) class I or II moderate not including the cusps, and touching the outside part of the middle of dentin. Assignment period will be 4 years: Inclusion period 18 months with 2 years following (6-month, 1 year and 2 years checking) and 3 months for statistical analysis and publications process Estimation of the parameters associated with a failure of the restoration at 24 months will follow the FDI scores. The Secondary objectives are to evaluate the caries risk of isolated population thanks to Cambra application and estimate the concordance of the judgment of maintaining the restoration between the expert in-situ and experts based on the images remotely.

ELIGIBILITY:
Inclusion Criteria:

* Patient with 2 carious lesions (or multiple of 2) class I or II moderate not including the cusps, and touching the outside part of the middle of dentin
* Asymptomatic tooth or with a reversible pulp syndrome tooth
* Measured by pulp test (if not possible should not prevent the inclusion)
* Patient consultant in investigative testing center
* Patient of 18 to 70 years old
* Patient able to support care
* Patient able to understand care (no language barrier)
* Collect the informed consent signed after a period of reflection
* Be affiliated to a French social security scheme or recipient of such a regime
* Tooth with criteria for pulp vitality tests of pulp sensibility

Exclusion Criteria:

* Patient under guardianship
* Pregnant or breastfeeding
* Patient at risk for infectious endocarditis
* Patient with severe periodontal disease (Pocket depth ≥ 5mm and/or mobility IV)
* Patient with an allergy to one of the materials used in the study
* Patient with an allergy to local anesthesia
* Patient with risks of infectious endocarditis
* Non-cooperative patient
* Participate in another ongoing biomedical research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the International Dental Federation Score | Change from Baseline Score FDI at 2 years
  Score are numbered from 1 to 5 in ascending order of severity for aesthetic criteria (5 items), functional criteria (9 items) and biological criteria (6 items). The score will be used by the practionner making the restoration and by the remote expert to check the results and validate tele-dentistry evaluation.

SECONDARY OUTCOMES:
Validation of the caries risk assememt. | Change from Baseline caries risk assement at 2 years
  Caries assessment is based on CAMBRA application https://course.mycambra.com/ (Caries Management By Risk Assessment) score giving 3 levels of caries assessment : Low - Moderate - High.
The carious presence according to the ICDAS / ICCMS criteria using the Soprolife® camera | At each follow-up visit (T0, T6 months, T1year and T2years)
  ICCMS: caries prevalence measurement based on the ICDAS classification

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France